CLINICAL TRIAL: NCT01428453
Title: A Phase 2a Study to Evaluate the Effect of Rilapladib (SB-659032) on Biomarkers Related to the Pathogenesis and Progression of Alzheimer's Disease
Brief Title: A Phase 2a Study to Evaluate the Effect of Rilapladib (SB-659032) in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114458
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — rilapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 250mg rilapladib (Experimental): Experimental drug
  Interventions: Drug: 250mg rilapladib
- placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 250mg rilapladib — Experimental Drug
  Arms: 250mg rilapladib
Drug: placebo — Placebo comparator
  Arms: placebo

SUMMARY:
The study is designed to investigate the effects of rilapladib on biomarkers related to the Alzheimer's disease, and cognitive function.

DETAILED DESCRIPTION:
The study is in subjects with Alzheimer's disease and evidence of cerebrovascular disease (CVD) who are currently treated with an acetylcholinesterase inhibitor (AChEI) and/or memantine. The study is a randomized, double-blind, placebo controlled, parallel group, repeat dose design, in which subjects (up to 60 randomized subjects per arm) will receive oral placebo or rilapladib (250 mg), once daily for 24 weeks in addition to their stable background AD therapy consisting of an acetylcholinesterase inhibitor (AChEI) and/or memantine. Subjects will take 250mg of rilapladib or placebo once daily for a period of 24 weeks. The total duration of participation for each subject will be approximately 30 weeks comprising approximately 4 weeks screening, 24 weeks treatment and 2 weeks follow-up. From the time of randomization and throughout the treatment period subjects will attend visits after 1 week, 4 weeks and thereafter every 4 weeks until Week 24. A follow-up visit will occur approximately 2 weeks after the final dose of study medication. Cognitive assessments will be performed at the screening visit, at the randomization (baseline) visit and at weeks 12 and 24 of the treatment period. Cerebrospinal fluid (CSF) samples will be taken via lumbar puncture at baseline and Week 24 for biomarker analyses related to Alzheimer's disease. Blood samples will be collected throughout the study for pharmacokinetics and a range of biomarker analyses. A range of safety and tolerability assessments will also be performed (including vital signs, laboratory tests, eye examinations and ECGs).

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of possible Alzheimer's disease in accordance with the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria, with radiological (Magnetic Resonance Imaging [MRI] or Computed Tomography [CT]) evidence of significant cerebrovascular disease (CVD), assessed within the last 12 months
2. Male or female between 50 and 80 years of age inclusive, at the time of signing the informed consent.
3. Subject has a documented history of at least 6 months of ongoing Alzheimer's disease therapy (AChEIs and/or memantine) with stable dosing for at least the last 2 months (and with no intent to change for the duration of the study).
4. Mini-Mental Status Examination (MMSE) score between 20 and 26 at Screening.
5. Clinical Dementia Rating Scale (CDR) score of 0.5 or 1.0 at Screening.
6. A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea; or of child-bearing potential and agrees to use acceptable contraception methods
7. Subject has provided full written informed consent prior to the performance of any protocol-specified procedure; or if the subject is unable to provide informed consent due to cognitive status, the subject will provide assent and full written informed consent will be provided by a legally acceptable representative
8. The subject has a dedicated caregiver who is willing to supervise participation in the study
9. In the opinion of the investigator, the subject has the ability to comply with study procedures (cognitive and other testing) and is fluent in the language used for the administration of the cognitive tests.

Exclusion Criteria:

1. History and/or evidence of any other CNS disorder that could be interpreted as a cause of dementia: e.g. structural or developmental abnormality, epilepsy, infectious, degenerative or inflammatory/demyelinating CNS conditions such as, Parkinson's disease and frontotemporal dementia
2. History of significant psychiatric illness such as schizophrenia or bipolar affective disorder that in the opinion of the Investigator would interfere with participation in the study; major depressive disorder (according to DSM-IV) in the past year; current active depression requiring initiation of treatment (or is believed to account for substantial degree of cognitive impairment)
3. Evidence of the following disorders: current vitamin B12 deficiency, positive syphilis serology (unless neurosyphilis was ruled out) or active thyroid dysfunction (particularly suggestive of hypothyroidism), including abnormally high or low serum levels of thyroid stimulating hormone (TSH), where this is thought to be the cause of, or to contribute to the severity of the subject's dementia.
4. History of alcohol or other substance abuse, according to the DSM-IV criteria, or recent or remote history of the same if that could be a contributing factor to dementia.
5. History of intra cerebral haemorrhage due to any of the following causes: cerebral amyloid angiopathy, uncontrolled hypertension, cerebral arteriovenous malformation, coagulopathy, CNS vasculitis or any other condition that the investigator and/or medical monitor considers as a relevant risk factor for intracerebral haemorrhage
6. Recent (i.e.,<6 months from Screening Visit) cardiovascular event defined as:

   1. ST-elevation MI or non-ST-elevation MI, confirmed by cardiac enzyme elevation and ECG changes
   2. coronary revascularization (percutaneous coronary intervention or coronary artery bypass graft )
   3. stroke of any etiology
   4. resuscitated sudden death
   5. prior carotid surgery or stenting procedure
7. Poorly controlled hypertension despite lifestyle modifications and pharmacotherapy (either systolic blood pressure >160mmHg or diastolic blood pressure >110mmHg)
8. QTcB interval >450 msec; or QTcB > 480 msec in subjects with bundle branch block based on ECG assessment at the Screening visit.
9. HbA1c >12.0 at Screening, or uncontrolled diabetes in the opinion of the investigator.
10. History of glaucoma or any other findings in the baseline eye exam that, in the opinion of the investigator, would exclude the subject from participation in the study.
11. History of adult asthma (or reactive airway disease) manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s).
12. Previous history of anaphylaxis, severe allergic reaction or history of hypersensitivity to any of the components of the formulation.
13. Significant abnormalities on clinical chemistry, haematology or urinalysis at Screening, including clinically significant anaemia.
14. History of chronic viral hepatitis (including presence of B surface antigen or hepatitis C antibody), or other chronic hepatic disorders.
15. Abnormal Screening blood tests exceeding any of the limits defined below:

    1. Alanine transaminase (ALT) or aspartate transaminase (AST) >1.5 x the upper limit of normal (ULN)
    2. Alkaline phosphatase (AP) and bilirubin >1.5X ULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
    3. Calculated creatinine clearance < 30 ml/min (per Cockcroft & Gault) at Screening
16. Other clinically significant abnormality on physical (including neurological), laboratory or ECG examination that could be detrimental to the subject in the opinion of the Investigator or could compromise the integrity of the study.
17. Planned major surgery within the study period.
18. Use of systemic steroids or other immunosuppressants within the last 30 days prior to screening.
19. Current treatment with barbiturates, MAO inhibitors, butyrophenones, phenothiazines and other "conventional" antipsychotic within 30 days or 5 half-lives prior to Screening, whichever is longer.
20. Treatment with antidepressants, (other than MAO inhibitors), thyroid hormones, atypical antipsychotics (e.g. risperidone), benzodiazepines and other sedatives / hypnotics unless prescribed at a stable dose for at least 2 months prior to Screening. Note: Benzodiazepines or other sedatives/hypnotics (including antihistamines) with half-life less than 6 hours can be taken on a prn (as needed) basis but must not be taken within 5 half lives prior to cognitive testing.
21. Current treatment with known potent inhibitors of CYP3A4 (e.g. ketoconazole, rifampin, modafinil).
22. Current treatment with known potent Pgp inhibitors (itraconazole, ketoconazole, cyclosporin, loperamide, diltiazem, verapamil, spironolactone, quinidine, bepridil, quinine, carvedilol)
23. Cognitive tasks prescribed for cognitive rehabilitation and performed under medical supervision in the 6 months prior to screening and/or during study
24. Investigational medications or devices including symptomatic AD treatment during the 60 days prior to the Screening visit, or within 5 half-lives of use of the investigational drug prior to the Screening Visit, whichever is longer.
25. Participation in another investigational drug (with the exception of anti-amyloid monoclonal antibodies [mAbs]) or device study where subject was treated chronically (i.e. > 1 single dose) with a study agent intended to impact AD progression during the 12 months prior to the Screening visit.

    1. Subjects who participated in an investigational drug study that involved chronic dosing with a monoclonal antibody at any time in the past are excluded from this study, unless it is known that they received placebo during the previous study.
    2. Subjects who participated in previous single-dose studies of anti-amyloid mAbs will be permitted provided the subject's dose of the mAb is at least 5 half-lives removed; the subjects did not experience any moderate adverse events classified as possibly drug-related or any serious adverse event during that study; the subject did not drop out of the previous study (i.e. completed all safety assessments)
26. Subjects, who in the investigator's judgement, pose a significant suicide risk (e.g. history of suicidal behaviour in the last 6 months and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 2 months).
27. Subject or caregiver is an immediate family member or employee of the participating Investigator, any of the participating site staff or GSK staff.
28. Any contraindication to lumbar puncture or insertion of CSF catheter, including but not limited to

    1. Thrombocytopenia or other coagulation disorders (including subjects receiving coumarin-derived anti-coagulants or low-molecular-weight heparin).
    2. The presence of cutaneous or soft tissue infection overlying or adjacent to the site of lumbar puncture.
    3. Previous spinal surgery that could complicate access to the subarachnoid space.
    4. Suspicion of increased intracranial pressure due to a cerebral mass.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-10-01; Primary Completion 2013-02-04 (Actual); Study Completion 2013-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- GSK Investigational Site, Sofia, Bulgaria
- Canada (3):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Germany (10):
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Oldenburg in Holstein, Schleswig-Holstein
- Italy (5):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Verona, Veneto
- GSK Investigational Site, Lørenskog, Norway
- Spain (6):
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Maher-Edwards G, De'Ath J, Barnett C, Lavrov A, Lockhart A. A 24-week study to evaluate the effect of rilapladib on cognition and cerebrospinal fluid biomarkers of Alzheimer's disease. Alzheimers Dement (N Y). 2015 Jun 30;1(2):131-140. doi: 10.1016/j.trci.2015.06.003. eCollection 2015 Sep. PMID 29854933
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114458 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114458 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114458 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114458 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114458 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114458 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114458 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Alzheimer's disease (AD) were randomized to either rilapladib or placebo from October-2011 to February-2013. The study duration was approximately 30 weeks (screening: 4 weeks, treatment: 24 weeks and follow-up: 2 weeks).
Pre-assignment Details: Total of 170 participants were screened, of which 124 were randomized in 24 centres. Out of 124 participants, one was excluded from safety population due to randomization error. Out of 123 participants, 2 were excluded due to unavailability of post-baseline efficacy data. Intention to treat (ITT) population consisted of 121 participants.
Groups:
- Placebo Once Daily: Participants randomized to receive oral placebo tablet once daily following breakfast for a period of 24 weeks. In addition, to their stable background therapy consisting of an acetylcholinesterase inhibitor (AChEI) and/or memantine.
- Rilapladib 250 mg Once Daily: Participants randomized to receive oral rilapladib 250 milligrams (mg) tablet once daily following breakfast for a period of 24 weeks. In addition, to their stable background therapy consisting of an AChEI and/or memantine.
Period: Overall Study
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Started | 62 | 61
Completed | 56 | 52
Not Completed | 6 | 9
Not completed — Adverse Event | 2 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: The data for ITT population is presented and defined as participants who were randomized, received at least one dose of study medication and had at least one non-missing post Baseline efficacy assessment. One participant from each group was excluded from ITT population as no post-baseline efficacy data available and total ITT population was 121.
Groups:
- Placebo Once Daily: Participants randomized to receive oral placebo tablet once daily following breakfast for a period of 24 weeks. In addition to their stable background therapy consisting of an AChEI and/or memantine.
- Rilapladib 250 mg Once Daily: Participants randomized to receive oral rilapladib 250 mg tablet once daily following breakfast for a period of 24 weeks. In addition to their stable background therapy consisting of an AChEI and/or memantine.
- Total: Total of all reporting groups
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (5.40) | 72.9 (5.15) | 73.0 (5.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 33 | 28 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European Heritage | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 0) in Cerebral Spinal Fluid (CSF) Amyloid Beta Peptide (Abeta) 42 and Abeta40 at Week 24
Description: CSF Abeta biomarkers (Abeta42, Abeta40) were assessed at Baseline visit (Day 0) and Week 24 (Day 168). Change from Baseline in CSF Abeta42 and Abeta40 are summarized. Baseline and Week 24 study visits were taken place at approximately the same time of day in the morning (preferably between 08:00 and 12:00) to improve the reliability of CSF. Baseline value was defined as the latest Day 0 value. Change from Baseline was calculated as post-dose (Week 24) visit value minus Baseline value. The data is presented in for adjusted mean and standard error of adjusted mean.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanograms per Liter
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 53 | 48
Nanograms per Liter
  Abeta42 | -6.3 (18.10) | 33.6 (19.02)
  Abeta40 | -77.4 (181.33) | -327.7 (190.56)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; p = 0.133, ANCOVA; The analysis method was ANCOVA adjusted for Treatment, Baseline CSF Abeta1-42 and Age; Mean Difference (Net) = 39.8, 95% CI 2-sided [-12.4 to 92.0] — Comparison of CSF Abeta42 between placebo and rilapladib 250 mg
Statistical Analysis 2: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; p = 0.829, ANCOVA; The analysis method was ANCOVA adjusted for Treatment, Baseline CSF Abeta1-40 and Age; Mean Difference (Net) = -250.3, 95% CI 2-sided [-771.9 to 271.2], Standard Error of Mean 265.66 — Comparison of CSF Abeta40 between placebo and rilapladib 250 mg

2. Primary Outcome: Change From Baseline (Day 0) in CSF Abeta42/ Abeta40 Ratio at Week 24
Description: CSF Abeta biomarkers (Abeta42, Abeta40) were assessed at Baseline visit (Day 0) and Week 24 (Day 168). Change from Baseline in CSF Abeta42/Abeta40 ratio is summarized. Baseline and Week 24 study visits were taken place at approximately the same time of day in the morning (preferably between 08:00 and 12:00) to improve the reliability of CSF. Baseline value was defined as the latest Day 0 value. Change from Baseline was calculated as post-dose (Week 24) visit value minus Baseline value. The data is presented in for adjusted mean and standard error of adjusted mean.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 53 | 48
Ratio | 0.002 (0.0068) | 0.018 (0.0071)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.016, 95% CI 2-sided [-0.003 to 0.036] — The analysis method was ANCOVA adjusted for Treatment, Baseline CSF Ratio Abeta1-42/Abeta1-40 and Age

3. Primary Outcome: Change From Baseline (Day 0) in CSF Tau and Phosphorylated Tau (P-tau) Measures at Week 24
Description: CSF tau and P-tau were assessed at Baseline visit (Day 0) and Week 24 (Day 168). Change from Baseline in CSF tau and P-tau was summarized. Baseline and Week 24 study visits were taken place at approximately the same time of day in the morning (preferably between 08:00 and 12:00) to improve the reliability of CSF. Baseline value was defined as the latest Day 0 value. Change from Baseline was calculated as post-dose (Week 24) visit value minus Baseline value. The data is presented in for adjusted mean and standard error of adjusted mean.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanograms per Liter
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 52 | 47
Nanograms per Liter
  CSF tau: number analyzed (Participants) | 52 | 46
  CSF tau | 38.2 (29.98) | -18.8 (31.90)
  P-tau | 1.3 (1.67) | -1.7 (1.76)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; p = 0.902, ANCOVA; The analysis method was ANCOVA adjusted for Treatment, Baseline CSF tau and Age; Mean Difference (Net) = -57.1, 95% CI 2-sided [-144.5 to 30.3], Standard Error of Mean 44.40 — Comparison of CSF tau between placebo and rilapladib 250 mg
Statistical Analysis 2: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; p = 0.892, ANCOVA; The analysis method was ANCOVA adjusted for Treatment, Baseline CSF P-tau and Age; Mean Difference (Net) = -3.0, 95% CI 2-sided [-7.9 to 1.8], Standard Error of Mean 2.46 — Comparison of P-tau between placebo and rilapladib 250 mg

4. Primary Outcome: Change From Baseline (Day 0) in the Computerized Test Battery for Cognition (CogState) Battery Working Memory/Executive Function (WM/EF) Composite Score at Week 24
Description: The WM/EF composite score was comprised of 5 functional tests including 1) Controlled oral word association which measured language fluency, planning and working memory, 2) Category naming: It measures semantic fluency, planning and working memory, 3) One-back: This is a measure of working memory. 4) Trail B: This is a measure of motor speed, visual scanning, and visual-motor integration. This test required attention and cognitive flexibility. 5) Go No-Go task: This test evaluate accuracy and reaction time for each response. The composite score calculated by standardizing the total score: sum of all responses obtained from these 5 functional test by using the formula (Total score of ITT population at baseline - Total score at Week 24) /standard deviation of mean total mean score at baseline. The observed composite score ranged from minimum -1.474 and maximum 1.596. Lower score means better cognitive status. Change from Baseline was calculated as post-dose visit minus Baseline value.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed. The data is presented in for adjusted mean and standard error of adjusted mean.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 56 | 48
Scores on a scale | -0.150 (0.0501) | 0.016 (0.0538)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; p = 0.026, Mixed-Model Repeated Measures analysis — The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline Working Memory/Executive Function Composite Score, Treatment by Visit and Baseline Working Memory/Executive Function Composite Score by Visit; Mean Difference (Net) = 0.167, 95% CI 2-sided [0.021 to 0.313] — A positive treatment difference indicates benefit, relative to placebo

5. Secondary Outcome: Change From Baseline (Day 0) in CSF Albumin Quotients at Week 24
Description: CSF albumin quotient was assessed at Baseline visit (Day 0) and Week 24 (Day 168). Change from Baseline in albumin quotient is summarized. Baseline and Week 24 study visits were taken place at approximately the same time of day in the morning (preferably between 08:00 and 12:00) to improve the reliability of CSF. Baseline value was defined as the latest Day 0 value. Change from Baseline was calculated as post-dose (Week 24) visit value minus Baseline value. The data is presented in for adjusted mean and standard error of adjusted mean.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanograms per Liter
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 46 | 40
Nanograms per Liter | 0.11 (0.172) | -0.13 (0.184)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; p = 0.828, ANCOVA; The analysis method was ANCOVA adjusted for Treatment, Baseline CSF Albumin Quotient and Age; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.74 to 0.26], Standard Error of Mean 0.256

6. Secondary Outcome: Change From Baseline (Day 0) in Plasma Levels of Abeta42 and Abeta40 at Week 24
Description: Plasma Abeta biomarkers (Abeta42, Abeta40) were assessed at Baseline visit (Day 0) and Week 24 (Day 168). Change from Baseline in plasma Abeta42 and Abeta40 are summarized. Baseline value was defined as the latest Day 0 value. Change from Baseline was calculated as post-dose (Week 24) visit value minus Baseline value. The data is presented in for adjusted mean and standard error of adjusted mean.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanograms per Liter
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 51 | 47
Nanograms per Liter
  Abeta42 | 1.5 (0.90) | 0.2 (0.94)
  Abeta40 | 8.8 (3.91) | 9.7 (4.06)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; Mixed-Model Repeated Measures analysis; Mean Difference (Net) = -1.3, 95% CI 2-sided [-3.9 to 1.2] — Comparison of Abeta42 between placebo and rilapladib 250 mg. The analysis method for Plasma parameters was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline, Treatment by Visit, Baseline by Visit and Age
Statistical Analysis 2: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; Mixed-Model Repeated Measures analysis; Mean Difference (Net) = 1.0, 95% CI [-10.2 to 12.2] — Comparison of Abeta40 between placebo and rilapladib 250 mg. The analysis method for Plasma parameters was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline, Treatment by Visit, Baseline by Visit and Age

7. Secondary Outcome: Change From Baseline (Day 0) in Plasma Levels of Abeta42/Abeta40 Ratio at Week 24
Description: Plasma Abeta biomarkers (Abeta42, Abeta40) were assessed at Baseline visit (Day 0) and Week 24 (Day 168). Change from Baseline in plasma Abeta42/Abeta40 ratio is summarized. Baseline value was defined as the latest Day 0 value. Change from Baseline was calculated as post-dose (Week 24) visit value minus Baseline value. The data is presented in for adjusted mean and standard error of adjusted mean.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 51 | 47
Ratio | -0.010 (0.0045) | -0.012 (0.0047)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; Mixed-Model Repeated Measures analysis; Mean Difference (Net) = -0.003, 95% CI 2-sided [-0.016 to 0.010] — The analysis method for Plasma parameters was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline, Treatment by Visit, Baseline by Visit and Age

8. Secondary Outcome: Percentage Inhibition in Plasma Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Activity at Week 24
Description: Plasma Lp-PLA2 was assessed at Baseline visit (Day 0) and Week 24 (Day 168). Percentage inhibition in plasma Lp-PLA2 activity ratio is summarized. Percentage inhibition was calculated by dividing change from Baseline in plasma LpPLA2 by Baseline LpPLA2 multiplied by -100. Baseline value was defined as the latest Day 0 value. Change from Baseline was calculated as post-dose (Week 24) visit value minus Baseline value.
Time Frame: Baseline (Day 0) and Week 24
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Placebo Once Daily: Participants randomized to receive oral rilapladib 250 mg tablet once daily following breakfast for a period of 24 weeks. In addition to their stable background therapy consisting of an AChEI and/or memantine.
- Rilapladib 250 mg Once Daily: Participants randomized to receive oral placebo tablet once daily following breakfast for a period of 24 weeks. In addition to their stable background therapy consisting of an AChEI and/or memantine.
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 53 | 47
Percent change | -3.86 (30.228) | 83.59 (10.483)

9. Secondary Outcome: Change From Baseline (Day 0) in CogState Battery Overall Composite Score
Description: CogState battery overall composite score comprised of 8 functional tests 1) Controlled oral word association test measured language fluency, planning and working memory. 2) Category naming test measured semantic fluency, planning and working memory. 3) One-back test measured working memory. 4) Trail B test measured motor speed, visual scanning and visual-motor integration, required attention and cognitive flexibility. 5) Go No-Go task evaluated accuracy and reaction time for each response. 6) International shopping list immediate and delayed recall tests measured episodic memory. 7) Identification task test assessed visual attention. 8) Trail A test measured psychomotor speed and attention. Composite score= total score (sum of all responses from 8 functional test) by formula (Total score at baseline - Week 24) / SD of total score at baseline. Score ranged: -1.070 to 0.907. Lower score indicated the better cognitive status. Change from Baseline= post-dose visit minus Baseline value
Time Frame: Baseline (Day 0) and Week 12 (Day 84), Week 24 (Day 168)
Population: ITT Population. Only those participants available at the specified time points were analyzed. The data is presented in for adjusted mean and standard error of adjusted mean.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 53 | 53
Scores on a scale
  Week 12: number analyzed (Participants) | 52 | 53
  Week 12 | 0.013 (0.0438) | -0.054 (0.0444)
  Week 24: number analyzed (Participants) | 53 | 48
  Week 24 | -0.121 (0.0445) | 0.017 (0.0466)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; Mixed-Model Repeated Measures analysis; Mean Difference (Net) = -0.067, 95% CI 2-sided [-0.191 to 0.057] — The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline Score, Treatment by Visit and Baseline Score by Visit. A positive treatment difference indicates benefit, relative to placebo. placebo
Statistical Analysis 2: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; p = 0.982, Mixed-Model Repeated Measures analysis — The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline Overall Composite Score, Treatment by Visit and Baseline Overall Composite Score by Visit; The probability (effect size) for change from Baseline in CogState battery overall composite score >0 is presented; Mean Difference (Net) = 0.138, 95% CI 2-sided [0.010 to 0.267] — A positive treatment difference indicates benefit, relative to placebo. Comparison of overall composite score between placebo and rilapladib 250 mg at Week 24

10. Secondary Outcome: Change From Baseline (Day 0) in CogState Battery Attention Composite Score
Description: CogState battery attention composite score comprised of 2 functional tests including 1) Identification task test assessed visual attention and 2) Trail A test measured psychomotor speed and attention. Composite score calculated by standardizing the total score (sum of all responses from 2 functional test) by formula (Total score at baseline - Week 24) / SD of total score at baseline. The observed composite score ranged from minimum -1.756 and maximum 1.330. Higher score indicated the better attention. Baseline value was defined as the latest Day 0 value and Change from Baseline was calculated as post-dose visit minus Baseline value
Time Frame: Baseline (Day 0) and Week 12 (Day 84), Week 24 (Day 168)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Once Daily | Rilapladib 250 mg Once Daily
Number analyzed (Participants) | 55 | 52
Scores on a scale
  Week 12: number analyzed (Participants) | 53 | 52
  Week 12 | -0.062 (0.0684) | -0.125 (0.0693)
  Week 24: number analyzed (Participants) | 55 | 48
  Week 24 | -0.089 (0.0686) | -0.019 (0.0729)
Statistical Analysis 1: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; Mixed-Model Repeated Measures analysis; The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline Score, Treatment by Visit and Baseline Score by Visit; Mean Difference (Net) = -0.063, 95% CI 2-sided [-0.257 to 0.130] — Comparison of attention composite score between placebo and rilapladib 250 mg at Week 12. A positive treatment difference indicates benefit, relative to placebo
Statistical Analysis 2: Comparison: Placebo Once Daily vs Rilapladib 250 mg Once Daily; Test type: Superiority or Other; Mixed-Model Repeated Measures analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Net) = 0.070, 95% CI 2-sided [-0.130 to 0.269] — Comparison of attention composite score between placebo and rilapladib 250 mg at Week 24. A positive treatment difference indicates benefit, relative to placebo

ADVERSE EVENTS:
Time Frame: Serious Adverse Event (SAE) and non-SAE were reported for treatment period only (up to Week 24).
Description: The safety population was used and defined as consisting of all participants who were randomized and received at least one dose of double-blind medication.
Groups:
- Rilapladib 250mg Once Daily: Participants randomized to receive oral rilapladib 250 mg tablet once daily following breakfast for a period of 24 weeks. In addition to their stable background therapy consisting of an AChEI and/or memantine.
Arm/Group | Placebo Once Daily | Rilapladib 250mg Once Daily
All-Cause Mortality (participants affected / at risk) | 1/62 | 1/61
Serious Adverse Events (participants affected / at risk) | 5/62 | 8/61
Other Adverse Events (participants affected / at risk) | 23/62 | 16/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Once Daily (N=62) | Rilapladib 250mg Once Daily (N=61)
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Complex partial seizures (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Once Daily (N=62) | Rilapladib 250mg Once Daily (N=61)
Headache (Nervous system disorders) | 10 (10) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (9) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 4 (6) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.